CLINICAL TRIAL: NCT06637566
Title: Effects Of Brandt Daroff Exercises With Cawthorne Cooksey Exercises On Balance, Dizziness And Functional Parameters In Older Adults With Vertigo
Brief Title: Effects of Brandt Daroff Exercises in Older Adults With Vertigo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0207
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vertigo
Keywords: Vertigo,; balance; functional parameters; dizziness,
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): They receive brandt daroff exercises with cawthorne cooksey exercises.
  Interventions: Other: Brandt Daroff exercises along with Cawthorne Cooksey exercises
- Control Group (Other): They receive brandt daroff exercises only.
  Interventions: Other: Brandt Daroff exercises

INTERVENTIONS:
Other: Brandt Daroff exercises along with Cawthorne Cooksey exercises — Brandt Daroff exercises along with Cawthorne Cooksey exercises. The Cawthorne Cooksey exercises include eye and head movements, coordination of eye and head movements (visual-vestibular interaction), postural control exercises, and progressively more difficult balance tasks (eyes open, eyes closed, large base support, uneven base support, while walking, in high visual or noisy environments). Exercises should be done three times a day, with 5 repetitions of each. The exercises will be performed in three sessions per week with 60 minutes each session for eight weeks. The cawthorne Cooksey exercises includes the following:
  A: Eye and head movement
  B: Head and body movement, sitting down:
  C: Standing up exercises:
  Arms: Experimental Group
Other: Brandt Daroff exercises — brandt daroff exercises without cawthorne Cooksey exercises. To begin the Brandt-daroff exercise, the patient will sit and swivel the head 45 degrees to one side (left), then instantly lie down on the other shoulder (right). The patient should be instructed to maintain this posture for 30 seconds or until the vertigo subsides. The patient then gradually returns to the starting position, maintaining the left ear rotation until sat upright. Following the same 30 second time limits, the patient turns his head in the opposite way (right) and rests down on the opposite shoulder (left). These exercises will be instructed to perform at home for 3 sets (morning, afternoon and evening) with 5 repetitions approximately for 30 minutes in each session for five weeks
  Arms: Control Group

SUMMARY:
Vertigo is among the most prevalent disorder in older adults around the world leads to dizziness and balance problems resulting in decreased quality of life. Brandt daroff exercises can accelerate vertigo recovery and prevent recurrence without taking drugs. Cawthorne Cooksey first presented vestibular exercises to improve neurophysiological habituation, improves balance in the elderly. This study aims to determine the effects of brandt daroff exercises with cawthorne cooksey exercises on balance, dizziness and functional parameters in older adults with vertigo.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Participants will be selected by non-probability convenience sampling technique, thirty two vertigo patients meeting the inclusion criteria will be randomly allocated into two equal groups (experimental and control) by online randomizer tool. The experimental group will receive brandt daroff exercises with cawthorne cooksey exercises and the control group will receive brandt daroff exercises alone. Treatment session of 60 min will be given 3 times a week for 6 weeks. The following assessment tool will be used Visual Analogue Scale and Dizziness Handicap Inventory for vertigo symptom severity, Berg Balance scale and Tinetti POMA for assessment of balance, Functional Independence Measure and IADL Tool for assessment of functional parameters. Assessment will be done at baseline and after 6 week. The data will be analyzed using SPPS software version. 25.

ELIGIBILITY:
Inclusion Criteria:

* Older adults 65or above.
* Both Male and Female.
* Symptoms suggested vertigo, confirmed by neurologist.
* Accepted to participate in study.
* DHI Scale: 36-42 (moderate handicap).

Exclusion Criteria:

* Patients having balance issues other than dizziness and vertigo.
* Middle or external ear diseases.
* Cerebrovascular diseases.
* Feet injuries including severe bruises, ulcers, open wounds or recent burns.
* Neck pain and cervical spine disease.
* History of serious musculoskeletal disease (arthritis, Alzheimer's disease, intervertebral disc degeneration).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory: | 6 weeks
  Dizziness Handicap Inventory (DHI) Scale is used for assessment of dizziness. DHI is 25-item self-report questionnaire that measures the impact of dizziness on a person's daily life and use as screening as well as outcome measuring tool in vertigo patients. Each item on the DHI is scored on a 0 to 4 scale, with 0 meaning "no problem" and 4 meaning "severe problem." It is a widely used tool in clinical practice to assess the severity of dizziness and its effect on a person's functional, emotional, and physical well-being. DHI has been found to have 75% sensitivity. The DHI Scale has been found to have high test-retest reliability (icc0.92) and moderate construct validity (Pearson's correlation coefficient 0.47). It is a self-report questionnaire so no special equipment is required to perform it.
Tinetti Performance Oriented Mobolity Assessment | 6 weeks
  Tinneti POMA (performance oriented mobility assessment) is a reliable tool use for assessment of balance and gait in older adults. The test and retest values for the POMA-T, POMA-B, POMA-G all varied between (0.72) and (0.86). The inter-rater reliability values all varied between (0.80) and (0.93). This test has a sensitivity of 70% and a specificity of 52%. It is a 17-item test that takes about 15 minutes to complete. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totaling 28.
  Equipment Required: A hard armless chair, A stopwatch, A 15 feet even and uniform walkway.
Lawton Instrumental Activities of Daily Living (IADL) Scale | 6 weeks
  The Lawton Instrumental Activities of Daily Living (IADL) Scale is used to evaluate independent living skills. The instrument is most useful for identifying how a person is functioning and identifying improvement or deterioration over time. The scale measures eight domains of function including food preparation, housekeeping, laundering. Individuals are scored according to their highest level of functioning in that category.
  A summary score ranges from 0(low function, dependent) to 8(high function, independent). Inter-rater reliability was established at.85. Administration time is10-15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Mphil, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Joharabad, Jauharabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixido M, Casserly R, Melley LE. Lateral Modified Brandt-Daroff Exercises: A Novel Home Treatment Technique for Horizontal Canal BPPV. J Int Adv Otol. 2021 Jan;17(1):52-57. doi: 10.5152/iao.2020.9452. PMID 33605222
- [Background] Zamyslowska-Szmytke E, Politanski P, Jozefowicz-Korczynska M. Dizziness Handicap Inventory in Clinical Evaluation of Dizzy Patients. Int J Environ Res Public Health. 2021 Feb 24;18(5):2210. doi: 10.3390/ijerph18052210. PMID 33668099